CLINICAL TRIAL: NCT00932854
Title: A Clinical tRial of Endobronchial Ultrasound for the Diagnosis of Isolated MEDiastinal lymphadenopathY (REMEDY)
Brief Title: A Clinical tRial of Endobronchial Ultrasound for the Diagnosis of MEDiastinal lymphadenopathY (REMEDY)
Acronym: REMEDY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Sam Janes, Reader in Respiratory Medicine, University College London Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REMEDY 09/0090
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Isolated Mediastinal Lymphadenopathy; Sarcoidosis; Tuberculosis; Lung Cancer; Lymphoma
Keywords: Mediastinal lymphadenopathy; EBUS; Bronchoscopy; Sarcoidosis
MeSH Terms: conditions — Sarcoidosis; Tuberculosis; Lung Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EBUS (Experimental): All patients in the trial will undergo EBUS for the diagnosis of isolated mediastinal lymphadenopathy. If this investigation is negative then the patient will be referred for mediastinoscopy.
  Interventions: Procedure: EBUS

INTERVENTIONS:
Procedure: EBUS — Endobronchial ultrasound guided transbronchial needle aspiration will be performed under conscious sedation and as an outpatient procedure. Additional bronchoscopy, transbronchial biopsies and bronchoalveolar lavage will be performed at the investigator's discretion.
  Other Names: EBUS-TBNA; EBUS-FNA

SUMMARY:
Enlarged glands in the chest (mediastinal lymphadenopathy) is a common problem and may have a variety of different causes. In the past an operation (mediastinoscopy) was required to diagnose the glands. Endobronchial ultrasound (EBUS) is a new procedure that may be able to diagnose these glands without the need for mediastinoscopy. The REMEDY trial aims to examine whether EBUS can reduce the number of mediastinoscopies and healthcare costs in patients with enlarged glands in the chest.

DETAILED DESCRIPTION:
Although the literature is replete with data on the utility of Endobronchial Ultrasound for lung cancer, there are very few data available on its role in the diagnosis of isolated mediastinal lymphadenopathy due to other causes such as sarcoid, tuberculosis or lymphoma. The REMEDY trial aims to evaluate the accuracy of EBUS in this setting and assess any reduction in the number of mediastinoscopies and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with undiagnosed mediastinal lymphadenopathy (>1cm in short axis) on CT or PET-CT scan for whom pathological evaluation is clinically indicated.

Exclusion Criteria:

* Patients without informed consent, those with anterior mediastinal lesions or with contra-indications to EBUS or mediastinoscopy will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Number of mediastinoscopies prevented and healthcare costs | At diagnosis

SECONDARY OUTCOMES:
Length of hospital stay | At diagnosis
Sensitivity and false negative rate of endobronchial ultrasound | At study completion

CONTACTS AND LOCATIONS:
Overall Officials: Sam Janes, MD PhD, Principal Investigator — University College, London; Neal Navani, MD, Study Director — Univeristy College London
Locations (1):
- University College London Hospital, London, London, United Kingdom

REFERENCES:
- [Derived] Navani N, Lawrence DR, Kolvekar S, Hayward M, McAsey D, Kocjan G, Falzon M, Capitanio A, Shaw P, Morris S, Omar RZ, Janes SM; REMEDY Trial Investigators. Endobronchial ultrasound-guided transbronchial needle aspiration prevents mediastinoscopies in the diagnosis of isolated mediastinal lymphadenopathy: a prospective trial. Am J Respir Crit Care Med. 2012 Aug 1;186(3):255-60. doi: 10.1164/rccm.201203-0393OC. Epub 2012 May 31. PMID 22652031